CLINICAL TRIAL: NCT05267938
Title: Microneedle Pretreatment as a Strategy to Improve the Effectiveness of Topical Anesthetics Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Texas Tech University (Other)
Responsible Party: Principal Investigator, Michelle Franz Montan Braga Leite, DDS, MSc, PhD, Principal Investigator, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 42926115.3.0000.5418
Record Dates: First submitted 2022-02-23; First posted 2022-03-07 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Oral Cavity Disease
Keywords: Microneedles; Oral Cavity; Transbuccal administration
MeSH Terms: conditions — Mouth Diseases | interventions — Anesthetics, Local; Therapeutics; Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant
Masking Description: Every volunteers has received bilateral pre-treatment with microneedles or the negative control in the palatal mucosa, in both sessions, which each session was 2 minutes of topical anesthetic or 5 minutes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microneedles (Experimental): Microneedles is with 750μm of height in order to prepare the palatal mucosa to receive the topical anesthetic
  Interventions: Drug: Topical Anesthetic; Drug: Local anesthetic
- patch flat (Sham Comparator): The same device as the microneedles but without microneedles
  Interventions: Drug: Topical Anesthetic; Drug: Local anesthetic

INTERVENTIONS:
Drug: Topical Anesthetic — The topical anesthetic used in this experimental is EMLA® after the pre-treatment of the palatal mucosa
  Other Names: treatment
Drug: Local anesthetic — After the pre-treatment with microneedles and the use of topical anesthetic, the needle and injection of local anesthetic was inserted and pain was evaluated
  Other Names: Lidocaine with epinephrine

SUMMARY:
A randomized, crossover, double-blind, two-sessions clinical trial with 30 male volunteers was performed to access pain of local anesthesia after using a topical anesthetic associated or not with prior application of microneedles to the palatal mucosa region

DETAILED DESCRIPTION:
A randomized, crossover, double-blind, two-sessions clinical trial with 30 male volunteers was performed by applying a microneedle patch and as a negative control the an identical patch but without microneedles sticking out and after the topical anesthetic was applied for in one session 2 minutes and the other session 5 minutes and the investigators evaluated the pain of needle introduction and the injection of the anesthetic.

The application force of the microneedles was standardized to 10N by an applicator composed of a 5 mL syringe and a spring. Pain and discomfort associated to the procedure was evaluated with a Visual Analogue Scale (VAS), in these two different moments, introduction of the needle and injection of the anesthetic.

ELIGIBILITY:
Inclusion Criteria:

- Healthy male

Exclusion Criteria:

* Volunteers were free from cardiac, hepatic, renal, pulmonary, neurological, gastrointestinal and haematological diseases, psychiatric disorders, smokers or alcoholic.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Pain sensitivity assessment by Visual Analogue Scale after the after puncture and injection of local anesthetic | 2 minutes or 5 minutes
  Microneedles or the negative control were used to prepare the palatal mucosa to receive the topical anesthetic, followed by the insertion of the needle and injection of the local anesthetic, evaluating whether the microneedles improve the effectiveness of the topical agent with a Visual Analogic Scale. The blind investigator, evaluated the values with a rule, the left far end mean 0, for no pain at all and the right far end mean 100 for maximum pain. Therefore, a higher score means a worse outcome,

CONTACTS AND LOCATIONS:
Locations (1):
- Michelle Franz Montan Braga Leite, Piracicaba, São Paulo, Brazil